CLINICAL TRIAL: NCT06538909
Title: Steps Against the Burden of Parkinson's Disease - StepuP
Acronym: StepuP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 0569-23-TLV
Record Dates: First submitted 2024-07-03; First posted 2024-08-06 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD with VR int. (Experimental): Parkinson's disease patients using Virtual reality intervention that include physical activity and cognitive
  Interventions: Device: VR

INTERVENTIONS:
Device: VR — Virtual reality that simulates obstacles on the road during walking
  Other Names: Virtual Reality

SUMMARY:
The goals of our StepuP project are:

1. To understand the kinematic and neural mechanisms underlying walking improvements due to treadmill training with and without VR-enabled gait adaptations in people with PD;
2. To assess to what extent improvements in walking due to treadmill training, as measured in the laboratory, transfer to improvements in daily life mobility;
3. To understand the mechanisms underlying the transfer from improvements in walking to improvements in mobility in daily life in people with PD;
4. To understand for whom treadmill training improves walking characteristics in the laboratory and for whom it does not, and to understand for whom treadmill training improves mobility in daily life and for whom it does not.

ELIGIBILITY:
Inclusion Criteria:

Specific criteria for Parkinson's disease - PD

* Diagnosis of Parkinson's disease according to the MDS World Movement Disorders Society criteria Disease severity H&Y I-III
* Score section 3.10 (ability to walk) MDS-UPDRS 3.10 ≥ 1
* MoCA cognitive assessment > 15
* Stable cardiovascular condition, ability to perform aerobic activity at low to moderate intensity
* Without orthopedic diseases and other diseases that affect the quality of walking, at the decision of the researcher.

Exclusion Criteria:

* Moderate or severe depression (BDI-II ≥18)
* Orthopedic diseases and other diseases that affect the quality of walking, at the decision of the researcher

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
motion capture | 13 months
  Kinematic data will be collected using a Qualisys or Vicon motion capture system at a sampling frequency of 100 Hz.
describe brain activity by EEG cap | 13 months
  EEG recordings will be made using a 64-channel or 128 channel EEG cap
describe muscles activity by EMG electrodes | 13 months
  Bipolar EMG electrodes will be placed on the leg muscles. EMG data will be recorded at a sample frequency available for each system around 2000 Hz.

SECONDARY OUTCOMES:
clinical trial TUG | 13 months
  standard time-up-and-go test
clinical trial walk test | 13 months
  2-minute walk test
clinical trial MiniBESTest | 13 months
  balance and fall risk
mGES questionnaire | 13 months
  modified gait efficacy scale
FES-i questionnaire | 13 months
  Short falls efficacy scale international FES-i
FACIT-F questionnaire | 13 months
  fatigue
EQ-5D questionnaire | 13 months
  health-related quality of life
Frailty questionnaire | 13 months
  Frailty index for physical activity
Fall questionnaires | 13 months
  Fall events (occurrence and frequency) and fall related injuries. (twelve-month retrospective during T0 and during the duration of the trail
MDS-UPDRS test | 13 months
  MDS-UPDRS
NFOGQ questionnaires | 13 months
  NFOGQ
aids questionnaires | 13 months
  Use of mobility aids
cognition questionnaires | 13 months
  MoCA and trail making test for cognition
Demographics questionnaire ( descriptive measures) | 13 months
  General descriptive measures : Year of birth, gender, height, weight, shoe size, education, employment, living arrangement, smoking history and alcohol consumption.
Fracture history questionnaire | 13 months
  Fracture history (number and type of fracture, twelve-month retrospective of T0)

IPD SHARING:
Plan to Share IPD: No